CLINICAL TRIAL: NCT06344130
Title: A Phase I Hypofractionation Trial of Re-irradiation in Good Prognosis Recurrent Glioblastoma
Brief Title: Hypofractionation Trial of Re-irradiation in Good Prognosis Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001859; 001859-C
Record Dates: First submitted 2024-04-02; First posted 2024-04-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-20

CONDITIONS: Astrocytoma; Glioma; Recurrent Glioblastoma
Keywords: Radiotherapy; Hypofractionation; Re-irradiation
MeSH Terms: conditions — Astrocytoma; Glioma; Glioblastoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1/Arm 1 (Experimental): Fraction size escalation of 3 planned re-irradiation dose levels.
  Interventions: Radiation: Radiation Therapy
- 2/Arm 2 (Experimental): MTD of re-irradiation dose.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation therapy will be administered via a linear accelerator using 6 megavoltage (MV) photons or greater.

SUMMARY:
Background:

Glioblastoma (GBM) is a cancer of the brain. Current survival rates for people with GBM are poor; survival ranges from 5.2 months to 39 months. Most tumors come back within months or years after treatment, and when they do, they are worse: Overall survival drops to less than 10 months. No standard treatment exists for people whose GBM has returned after radiation therapy.

Objective:

To find a safe schedule for using radiation to treat GBM tumors that returned after initial radiation treatment.

Eligibility:

People aged 18 years and older with grade 4 GBM that returned after initial radiation treatment.

Design:

Participants will be screened. They will have a physical exam with blood tests. A sample of tumor tissue may be collected.

Participants will undergo re-irradiation planning: They will wear a plastic mask over their head during imaging scans. These scans will pinpoint the exact location of the tumor. This spot will be the target of the radiation treatments.

Participants will undergo radiation treatment 4 times per week. Some people will have this treatment for 3 weeks, some for 2 weeks, and some for 1 week. Blood tests and other exams will be repeated at each visit.

Participants will complete questionnaires about their physical and mental health. They will answer these questions before starting radiation treatment; once a week during treatment; and at intervals for up to 3 years after treatment ends.

Participants will have follow-up visits 1 month after treatment and then every 2 months for 6 months. Follow-up clinic visits will continue up to 3 years. Follow-ups by phone or email will continue an additional 2 years.

DETAILED DESCRIPTION:
Background:

* Although survival of glioblastoma (GBM) has improved using standard of care chemoradiation, outcomes are still poor. Most patients will recur within months to years, in or adjacent to their previous treatment field.
* There is no consensus standard of care for patients with recurrent GBM. Re-resection is recommended, if possible, to improve symptoms and decrease tumor volume. However, this treatment option is possible only in a minority of patients, and for these patients re-irradiation has emerged as a possible treatment.
* Modern radiation therapy (RT) techniques allow delivery of reirradiation while minimizing the dose to previously treated organs at risk (OAR) within the radiation field.
* Data from a recently completed clinical trial at our center (16-C-0081, NCT02709226) suggests that the Maximum Tolerated Dose (MTD) of re-irradiation in 350 cGy fractions is 4200 cGy.

Objective:

-To determine the maximum tolerated dosage of daily re-irradiation in participants with recurrent Grade 4 gliomas

Eligibility:

* A histologic diagnosis of GBM, gliosarcoma, or transformation, from a lower grade to a grade 4 brain tumor.
* Previous glioma irradiation to curative-intent doses.
* Age >= 18.
* Karnofsky performance scale (KPS) >= 70.

Design:

* This is a single center phase I trial using a '3 plus 3' design and a three (3) dose level hypofractionation schema to enroll a maximum of 21 evaluable participants.
* Prior to radiation therapy, participants will undergo laboratory evaluations, magnetic resonance imaging (MRI), and a treatment planning computed tomography (CT).
* RT will be administered daily 4 days a week for 1, 2, or 3 weeks in the Radiation Oncology Branch, NCI, at NIH. Radiation will be delivered on consecutive days, 4 fractions per week via a linear accelerator using 6 megavoltage (MV) photons or greater.
* Follow-up visits following RT are planned at 1 month, every 2 months for years 1-2, and every 3 months for year 3. These visits will be stopped earlier in case of progression. After progression or 3 years of follow-up, participants will be followed remotely for survival

until 5 years after treatment completion.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologic diagnosis of primary glioblastoma or gliosarcoma of the brain, or secondary glioblastoma of the brain due to transformation from a lower grade to a grade 4 tumor.
* Age >= 18.
* KPS >= 70%.
* Previous tumor irradiation to curative-intent doses.
* Radiation dose constraints must be achievable based on assessment with MRI and treatment planning CT.
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) >= 1,000/microL
  * Platelets >= 100,000/microL
  * Coagulation: Prothrombin time (PT) / Partial thromboplastin time (PTT) within institutional normal range.
  * Total and direct bilirubin < 2 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) < 2 x institutional ULN
  * Alanine transaminase (ALT) < 2 x institutional ULN
  * Serum creatinine < 1.5 mg/dL
  * Serum albumin >= 0.75 x institutional normal range
* Individuals of child-bearing potential (IOCBP) and individuals who can father children must agree to use effective contraception (barrier, hormonal, intrauterine device, surgical sterilization, abstinence) from study entry and through 6 months after the last study treatment (restricted period). Individuals who can father children must not freeze or donate sperm within the same period.
* Nursing participants must be willing to discontinue nursing from study treatment initiation through 6 months after the last study treatment.
* The ability of a participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Recent systemic therapy prior to the initiation of the study therapy as follows:

  * Bevacizumab used for reasons other than tumor progression or symptomatic management within 2 weeks.
  * Temozolomide within 2 weeks.
  * Cytotoxic chemotherapy within 3 weeks.
  * Any investigational agents within 2 weeks.
* Participants who are unable to undergo MRI evaluation or receive gadolinium contrast for any reason.
* Any prior therapy after surgical re-resection or biopsy within 2 weeks prior to the initiation of the study therapy.
* Requiring radiation therapy within 12 months prior to the initiation of study therapy.
* History of prior therapy with Novacure TTF, Gliadel wafers, or GammaTile therapy.
* Positive beta-human chorionic gonadotropin (HCG) pregnancy test performed in individuals of childbearing potential at screening.
* Participants with known or suspected radiation sensitivity syndromes.
* Uncontrolled intercurrent illness evaluated by medical history and physical exam that are not stable and would potentially increase the risk to the participant.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD of daily re-irradiation in participants with recurrent grade 4 gliomas | DLT period (28 days)
  The number of participants experiencing DLTs within the DLT period will be reported for each hypofractionation schema. The MTD will be identified, and the proportion of participants treated with the MTD experiencing DLT will be reported.

SECONDARY OUTCOMES:
Progression free survival | Baseline, 30 day safety follow up visit, every 2 months for 2 years, every 3 months for 3rd year, or until progression
  Time to progression is defined as the interval from the initiation of treatment on protocol to progression or death. Estimates of the median time to progression and of the proportion of participants experiencing progression by 3 years or dying by 5 years will be obtained.
Overall survival | Treatment and follow up
  Overall survival is defined as the interval from initiation of treatment on protocol to the death. Estimates of the median time to overall survival will be obtained.
Compliance and feasibility of administering PRO in this participant population | Baseline through 3 years post radiation therapy.
  Patient reported outcome forms will be checked versus the timing schedule and considered valid if they fall within the scheduled assessment window. Compliance rates, namely the number of received valid forms over the number of expected forms will be reported.
Tolerability of treatment by assessing adverse events, cognitive function, physical function, and side effect bother | First radiation treatment administration through 6 months after the last day of radiation. Beyond 6 months after radiation, only adverse events which are serious and related to radiation need to be recorded.
  Tolerability of treatment will be assessed by determining the frequency of adverse events among treated participants and reporting the results by maximum grade of event and type of toxicity noted.
Longitudinally describe and evaluate disease and treatment-related symptom severity and interference with daily activities | Baseline through 3 years post radiation therapy.
  Longitudinal changes in perceived cognition, disease and treatment-related symptom severity, and interference with daily activities will be evaluated and described. The proportion of participants rating their symptoms as mild , moderate, or severe for individual symptoms will be reported.
Meaningful change in disease and treatment-related symptoms by using anchors | Baseline through 3 years post radiation therapy.
  Meaningful change will be determined through both clinician-rated (Karnofsky) and participant-rated (PGI-Severity, PGI-Change) anchors from the MD Anderson Symptom Inventory for Brain Tumors and Montreal Cognitive Assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter GK Mathen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers after the completion of the primary endpoint.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001859-C.html